CLINICAL TRIAL: NCT06810011
Title: EyeMatics - Eye Diseases "Treated" with Interoperable Medical Informatics
Brief Title: Eye Diseases "Treated" with Interoperable Medical Informatics
Acronym: EyeMatics
Status: Recruiting | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: University Medicine Greifswald (Other); University Medical Center Mainz (Other); University Hospital, Aachen (Other); Klinikum Chemnitz gGmbH (Other); Technische UniversitÃ¤t Dresden (Unknown); University of Leipzig (Other); University Hospital Tuebingen (Other); Deutsche Ophthalmologische Gesellschaft e.V. (Unknown); Pro Retina Deutschland e.V. (Unknown)
Responsible Party: Principal Investigator, Nicole Eter, Univ.-Prof. Dr. med. Nicole Eter, University Hospital Muenster
Other Study IDs: 01ZZ2319A-I; 01ZZ2319A-I (Other Grant/Funding Number: Federal Ministry of Education and Research)
Record Dates: First submitted 2024-12-12; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Intravitreal Injections
Keywords: Artificial intelligence; Core dataset; Intraviteal Injection; Medical Informatics; Data exchange

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The overarching goal of EyeMatics is to promote an interoperable, sustainable infrastructure for the integration and sharing of data from clinical research to improve personalized medicine in ophthalmology. To achieve this, EyeMatics bundles the expertise and preliminary work of the four consortia of the Medical Informatics Initiative (MII) and the ophthalmological centers of excellence in Germany. The perspective and concerns of patients will be strongly incorporated into the project work through close cooperation with patient representatives and the inclusion of patient feedback on quality of life and treatment success.

EyeMatics aims to improve the understanding of the therapeutic success of eye diseases that are usually treated with intravitreal surgical medication (IVOM). To this end, an exemplary analysis platform for "real" clinical data will be provided and a dashboard for data visualization and analysis will be developed as a web application. The dashboard is to be introduced at all participating hospital sites for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* OPS code: "5-156.9 Injection of drugs into the posterior segment of the eye"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving intravitreal injections at the study centers with signed Broad Consent (Consent of the Medical Informatics Initiative Germany).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Medical success | with every treatment or controll-visit within 12, 24 and 36 months
  changes in visual acuity during the course of treatment

SECONDARY OUTCOMES:
Treatment latency period: | from indication to treatment begin (Depending on the treatment regimen, assessed up to 6 months)
  latency period within the treatment and monitoring cycle as days between the indication/OCT examination and the implementation of IVOM treatment
Treatment and monitoring frequency | during the procedure
  Considered for the injection upload phase and for the first 12, 24 and 36 months of treatment. The number of injections is evaluated at patient level as a quality indicator and for the various treatment regimens, indications and clinical centers.
Treatment adherence | during the procedure
  Non-adherence to treatment is defined as those patients who did not receive any control or therapy without a planned treatment/control gap of 3 months.
Treatment persistence | during the procedure
  Treatment non-persistence is defined as the number of patients who received no further monitoring or treatment for a period of at least 6 months and did not resume treatment at the time of analysis.
Patient-relevant outcomes (PROMs) | every 6 months within 12, 24 and 36 months
  intravitreal injection specific PROM-questionnaire, including aspects of visual quality of life, socio-emotional quality of life, therapy and therapy environment, process quality, internal quality management, knowledge of the disease and pain

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Universitätsklinikum Aachen, AöR, Aachen
  - Universitätsmedizin Greifswald, Greifswald
  - Universität Leipzig, Leipzig
  - Universität Münster, Münster
  - Universitätsklinikum Tübingen, Tübingen

REFERENCES:
- [Background] Holtrup L, Varghese J, Schuster AK, Poschkamp B, Hampf C, Waltemath D, Wahle L, Lipprandt M, Merle DA, Berens P, Kohlbacher O, Kakkassery V, Bartos M, Ziemssen F, Wendt T, Hoffmann K; EyeMatics Study Group; Eter N. [EyeMatics-Multicenter data evaluation of real-world data with interoperable medical informatics]. Ophthalmologie. 2025 Apr;122(4):270-277. doi: 10.1007/s00347-024-02135-0. Epub 2024 Nov 14. German. PMID 39542916